CLINICAL TRIAL: NCT05620992
Title: Evaluation of Right Ventricular Function Post Mitral Valve Operations in Patients With Pulmonary Hypertension.
Brief Title: Evaluation of Right Ventricular Function Post Mitral Valve Operations
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Ali Mohammad Abdelbakey, Resident, Assiut University
Other Study IDs: Right ventricular function
Record Dates: First submitted 2022-11-12; First posted 2022-11-17 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Echocardiography 3 and 6 months post operative

SUMMARY:
We aim to determine the function of Right ventricle post mitral valve surgeries in patients with pulmonary hypertension using transthoracic echocardiography3- and 6-months post-operatively to detect the effect of mitral valve surgeries over the RV function whether improving, deteriorating, or not changing at all.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent mitral valve surgeries who also had pulmonary hypertension in the period between March 2019 and March 2022 in Assiut university heart hospital

Exclusion Criteria:

* Patients who underwent mitral valve surgeries with normal pulmonary pressure. Patients who had other valve surgeries besides mitral as aortic and/or tricuspid valve surgeries. Patients had mitral valve surgeries with other heart conditions that needed another intervention in the same session as CABG for IHD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Descriptive cross-sectional
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Right Ventricular function post mitral valve surgeries in patients with pulmonary hypertension | From March 2019 till March 2022
  to detect right ventricular function (ejection fraction percentage and/or TAPSE) through transthoracic echocardiography 3- and 6-months post operatively in patients who had mitral valve surgeries with pulmonary hypertension.

SECONDARY OUTCOMES:
Best mitral valve surgical modalities in patients with pulmonary hypertension | From March 2019 till March 2022
  to identify best surgical modalities for mitral valve diseased patients with pulmonary hypertension that lead to improvement of right ventricle function.

REFERENCES:
- [Background] Ho SY. Anatomy of the mitral valve. Heart. 2002 Nov;88 Suppl 4(Suppl 4):iv5-10. doi: 10.1136/heart.88.suppl_4.iv5. No abstract available. PMID 12369589
- [Background] Tokodi M, Nemeth E, Lakatos BK, Kispal E, Toser Z, Staub L, Racz K, Soltesz A, Szigeti S, Varga T, Gal J, Merkely B, Kovacs A. Right ventricular mechanical pattern in patients undergoing mitral valve surgery: a predictor of post-operative dysfunction? ESC Heart Fail. 2020 Jun;7(3):1246-1256. doi: 10.1002/ehf2.12682. Epub 2020 Mar 26. PMID 32220010
- [Background] Denault A, Deschamps A, Tardif JC, Lambert J, Perrault L. Pulmonary hypertension in cardiac surgery. Curr Cardiol Rev. 2010 Feb;6(1):1-14. doi: 10.2174/157340310790231671. PMID 21286273
- [Background] Estrada VH, Franco DL, Moreno AA, Gambasica JA, Nunez CC. Postoperative Right Ventricular Failure in Cardiac Surgery. Cardiol Res. 2016 Dec;7(6):185-195. doi: 10.14740/cr500e. Epub 2016 Dec 31. PMID 28197291
- [Background] Nagel E, Stuber M, Hess OM. Importance of the right ventricle in valvular heart disease. Eur Heart J. 1996 Jun;17(6):829-36. doi: 10.1093/oxfordjournals.eurheartj.a014963. PMID 8781821